CLINICAL TRIAL: NCT03447730
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacodynamics of SYNB1020 in Hepatic Insufficiency and Cirrhosis Patients
Brief Title: Safety, Tolerability and Pharmacodynamics of SYNB1020
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Interim futility analyses identified a lack of SYNB1020 efficacy.
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYNB1020-CP-002
Record Dates: First submitted 2018-02-16; First posted 2018-02-27 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 was open-label; Part 2 was double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: SYNB1020 (Experimental): Part 1 comprised a sentinel open-label cohort of subjects enrolled sequentially to receive SYNB1020, which was administered orally at a dose of 5 × 10^11 colony-forming units (CFU) 3 times daily (TID) given immediately after meals from Days 1 through 6.
  Interventions: Drug: SYNB1020
- Part 2: SYNB1020 (Experimental): Subjects randomized to receive SYNB1020 in Part 2 received SYNB1020 administered orally at a dose of 5 × 10^11 CFU TID given immediately after meals from Days 1 through 6.
  Interventions: Drug: SYNB1020
- Part 2: Placebo (Placebo Comparator): Subjects randomized to receive control in Part 2 received matching placebo (100 mL masking solution) administered orally TID given immediately after meals from Days 1 through 6.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SYNB1020 — SYNB1020 was supplied at a concentration of approximately 1 × 10^11 CFU/mL in a buffered solution in 5 mL cryovials with a nominal 5 mL fill volume, administered with 100 mL of masking buffer solution.
  Arms: Part 1: SYNB1020; Part 2: SYNB1020
Other: Placebo — Subjects received placebo orally in a chilled buffered solution (100 mL).
  Arms: Part 2: Placebo

SUMMARY:
This Phase 1b/2a, randomized, double-blind, placebo-controlled study was designed to evaluate the safety, tolerability, and pharmacodynamics of SYNB1020 in hepatic insufficiency and cirrhosis patients with hyperammonemia, with dosing of the investigational medicinal product (IMP) administered in an inpatient unit and subsequent outpatient follow-up for SYNB1020 clearance in two study parts.

DETAILED DESCRIPTION:
In Part 1, a sentinel open-label cohort of subjects with cirrhosis and Model for End-Stage Liver Disease (MELD) score <12 was admitted to an inpatient facility for a run-in diet, baseline assessments, IMP administration, safety monitoring, and collection of blood, urine, and stool samples for evaluation of safety, tolerability, and pharmacokinetic (PK) and pharmacodynamic (PD) evaluations. Subjects in Part 1 were enrolled sequentially to receive SYNB1020. Once the safety and tolerability were established in Part 1, enrollment was opened to subjects in Part 2.

Part 2 comprised a randomized, double-blind, placebo-controlled study in subjects with cirrhosis and hyperammonemia. Subjects were permitted to be pre-screened for eligibility based on medical history and a single fasting spot venous ammonia measurement. Eligible subjects with elevated fasting spot venous ammonia then underwent full screening within 7 days of pre-screening. Eligible subjects were admitted to an inpatient facility for a run-in diet and 24-hour ammonia profile, and those with an elevated 24-hour ammonia area under the curve (AUC) (>1.2 × the upper limit of normal [ULN]) proceeded with computer-generated randomization in a 1:1 ratio to receive either SYNB1020 or matching placebo. Randomization was followed by IMP administration, safety monitoring, and collection of blood, urine, and stool samples for PK and PD evaluations.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 to < 75 years
* Females must have been of non-childbearing potential
* Able and willing to complete informed consent process
* Available for and agreed to all study procedures
* Screening laboratory evaluations within defined acceptable limits or judged to be not clinically significant by the Investigator
* Diagnosis of chronic, stable, hepatic insufficiency with features of cirrhosis due to any etiology
* Evidence of elevated portal hypertension by either liver stiffness measurement, the presence of abdominal or esophageal varices, splenomegaly or ascites (Part 2 only)
* Elevated venous ammonia (Part 2 only)

Key Exclusion Criteria:

* Body mass index < 18.5 or ≥ 40 kg/m^2
* Administration or ingestion of an investigational drug within 8 weeks or 5 half-lives, whichever was longer, prior to screening or current enrollment in an investigational study
* Allergy to ranitidine or intolerance to any of the excipients (glycerol, CS Health Easy Fiber)
* Any condition, prescription medication or over-the-counter product that may possibly have affected absorption of medications or nutrients
* Dependence on drugs of abuse
* Apart from chronic liver disease, any acute or chronic medical, surgical, psychiatric, or social condition including history of cerebrovascular disease (stroke, transient ischemic attack) or dementia, or laboratory abnormality that may have increased the subject risk associated with study participation, compromised adherence to study procedures and requirements, confounded interpretation of the safety, kinetics, or PD results, and, in the judgment of the Investigator, made the subject inappropriate for enrollment
* Current or past hepatic encephalopathy of Grade 2 or higher requiring hospitalization
* Child-Turcotte-Pugh score > 9
* History of liver transplant

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Southern California Research Center, Coronado, California
  - Inland Empire Liver Foundation, Rialto, California
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Liver Institute, San Antonio, Texas
  - McGuire VA Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1: SYNB1020 | Part 2: SYNB1020 | Part 2: Placebo
Started | 6 | 9 | 8
Completed (Completed all 6 days of TID dosing) | 6 | 7 | 8
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of study treatment
Groups:
- Part 1: SYNB1020: Part 1 comprised a sentinel open-label cohort of subjects enrolled sequentially to receive SYNB1020, which was administered orally at a dose of 5 × 10^11 CFU TID given immediately after meals from Days 1 through 6.
- Total: Total of all reporting groups
Arm/Group | Part 1: SYNB1020 | Part 2: SYNB1020 | Part 2: Placebo | Total
Number analyzed (Participants) | 6 | 9 | 8 | 23
Age, Continuous [Median (Full Range); unit: years] | 54.5 [35.0 to 68.0] | 57.0 [38.0 to 74.0] | 59.5 [45.0 to 74.0] | 58.0 [35.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 7
  Male | 4 | 5 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 6 | 13
  Not Hispanic or Latino | 3 | 5 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 9 | 8 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, as follows: Grade 1 (mild/asymptomatic; no intervention); Grade 2 (moderate; minimal intervention); Grade 3 (severe/medically significant; hospitalization indicated; disabling); Grade 4 (life-threatening; urgent intervention required). Adverse events (AEs) were reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, and any other medically indicated assessments, including subject interviews, from the time informed consent was signed through the end of the safety follow-up period. AEs were considered to be treatment emergent adverse events (TEAEs) if they occurred or worsened in severity after the first dose of study treatment. TEAEs were considered treatment-related if relationship to study drug was possibly related, probably related, definitely related, or a missing relationship.
Time Frame: Up to 70 days
Population: All subjects who received at least 1 dose of SYNB1020 or placebo
Measure: Number; unit: participants
Arm/Group | Part 1: SYNB1020 | Part 2: SYNB1020 | Part 2: Placebo
Number analyzed (Participants) | 6 | 9 | 8
participants
  Any TEAE | 4 | 8 | 4
  Maximum TEAE severity Grade 1 | 3 | 3 | 1
  Maximum TEAE severity Grade 2 | 1 | 5 | 2
  Maximum TEAE severity Grade 3 | 0 | 0 | 1
  Treatment-related TEAE | 2 | 4 | 0
  TEAE leading to discontinuation | 0 | 2 | 0
  Treatment-related TEAE leading to discontinuation | 0 | 0 | 0
  Serious TEAE | 0 | 0 | 1
  Treatment-related Serious TEAE | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Clearance of SYNB1020 From Feces
Description: SYNB1020 transit through the gastrointestinal tract was measured with qualitative and quantitative polymerase chain reaction (PCR) fecal assays from fecal samples collected at baseline, daily during the dosing period (Days 1 through 6), at the time of discharge from the inpatient unit (Day 7), and at follow-up visits beginning 7±1 days after the last dose and continuing biweekly until a subject had a negative SYNB1020 fecal test. SYNB1020 clearance reflects a test value of below the limit of quantitation (BLQ) occurring after the indicated number of days following the last dose of study treatment.
Time Frame: Up to 65 days
Population: All subjects who received at least 1 dose of SYNB1020 or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: SYNB1020 | Part 2: SYNB1020 | Part 2: Placebo
Number analyzed (Participants) | 6 | 9 | 8
Participants
  Cleared by 25 days after last dose | 6 | 9 | 0
  SYNB1020 presence not detected | 0 | 0 | 8

3. Secondary Outcome: Daily Fasting Spot Venous Ammonia
Description: Fasting spot venous ammonia was collected at baseline (Day -2) and at the time of discharge from the inpatient unit (Day 7).
Time Frame: Up to 9 days
Population: All subjects who received at least 1 dose of SYNB1020 or placebo, completed the study, and were considered evaluable for analysis of pharmacodynamic data
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 1: SYNB1020 | Part 2: SYNB1020 | Part 2: Placebo
Number analyzed (Participants) | 6 | 7 | 8
μmol/L
  Baseline | 64.7 (25.00) | 82.0 (36.41) | 55.6 (18.18)
  End of Study/Day 7 | 62.3 (27.57) | 97.7 (58.79) | 67.9 (42.69)

ADVERSE EVENTS:
Time Frame: All AEs occurring from the time a subject signs informed consent through the safety follow-up period (i.e.,up to 70 days) were documented, regardless of the causal relationship to study drug. AEs that occurred or worsened in severity after the first dose of study treatment were considered treatment emergent (i.e., TEAEs).
Description: AE documentation included duration (onset and resolution dates), severity using the NCI CTCAE (version 4.03), assessment of causality, seriousness, and whether specific action or therapy was required. In summaries, preferred terms are counted only once per subject at the maximum reported grade.
Arm/Group | Part 1: SYNB1020 | Part 2: SYNB1020 | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 1/8
Other Adverse Events (participants affected / at risk) | 4/6 | 8/9 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: SYNB1020 (N=6) | Part 2: SYNB1020 (N=9) | Part 2: Placebo (N=8)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Severity Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: SYNB1020 (N=6) | Part 2: SYNB1020 (N=9) | Part 2: Placebo (N=8)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) — Maximum severity Grade 1
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) — Maximum severity Grade 2
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) — Maximum severity Grade 2
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) — Maximum severity Grade 2
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Maximum severity Grade 2
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Maximum severity Grade 2
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Maximum severity Grade 1
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) — Maximum severity Grade 2
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) — Maximum severity Grade 2
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) — Maximum severity Grade 2
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Maximum severity Grade 1
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Maximum severity Grade 1
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Maximum severity Grade 1
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Maximum severity Grade 2
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) — Maximum severity Grade 2
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Maximum severity Grade 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Maximum severity Grade 2
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Maximum severity Grade 1
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Maximum severity Grade 1

LIMITATIONS AND CAVEATS:
Interim futility analyses identified a lack of SYNB1020 efficacy (plasma ammonia AUC) compared with placebo, resulting in study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03447730/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03447730/SAP_000.pdf